CLINICAL TRIAL: NCT05838183
Title: Study on the Clinical Characteristics of Interstitial Lung Disease and Obstructive Sleep Apnea
Brief Title: Interstitial Lung Disease and Obstructive Sleep Apnea
Status: Recruiting | Type: Observational
Sponsor: Dan Liu (Other)
Responsible Party: Sponsor-Investigator, Dan Liu, Master of Medicine, attending physician, Tianjin Medical University General Hospital
Organization: Tianjin Medical University General Hospital (Other)
Other Study IDs: Dliu
Record Dates: First submitted 2023-04-10; First posted 2023-05-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: ILD OSA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Alveolar lavage fluid、Lung tissue、Blood samples or other samples

GROUPS / COHORTS (2):
- ILD with OSA group: ILD patient diagnosed with OSA by PSG. Bronchoscopy was performed to obtain alveolar lavage fluid in ILD patients and lung tissue was obtained for ROSE and mNGS in appropriate patients
  Interventions: Diagnostic Test: The relationship between imaging and ROSE and NGS
- ILD without OSA: ILD patients excluded OSA through PSG. Bronchoscopy was performed to obtain alveolar lavage fluid in ILD patients and lung tissue was obtained for ROSE and mNGS in appropriate patients
  Interventions: Diagnostic Test: The relationship between imaging and ROSE and NGS

INTERVENTIONS:
Diagnostic Test: The relationship between imaging and ROSE and NGS — The correlation between ROSE and NGS in imaging and bronchoscopy of ILD patients was observed
  Other Names: Association between the severity of OSA and biological specimen examination

SUMMARY:
Clinically, all patients with interstitial lung disease(ILD) were observed, and relevant clinical data were collected. Bronchoscopic specimens were collected according to the condition of the enrolled patients, and the rapid on site evaluation(ROSE) was evaluated, combined with the metagenomic next generation sequencing(mNGS) results of these patients. To observe the etiology and biological characteristics of exacerbation in patients with interstitial lung disease.

All patients undergo polysomnography (PSG) and drug-induced sleep endoscopy(DISE). The biological specimens was obtained for molecular biology or other tests.We detected ZNF331, Claudin1, Claudin2, Claudin3, Claudin4, and IL22 as biomarkers to differentiate the diagnostic efficiency of OSA in ILD, ILD+OSA, OSA, and Ctrl groups, respectively

ELIGIBILITY:
Inclusion criteria:

* over 18 years old and under 80 years old.
* Clinical diagnosis of interstitial lung disease or obstructive respiratory sleep apnea syndrome.
* Patient is conscious and capable of signing informed consent.
* The patient may wear a polysomnograph.

Exclusion criteria:

* malignant tumors.
* severe heart failure.
* uremia.
* autoimmune diseases.
* pulmonary embolism, and end-stage chronic obstructive pulmonary disease.
* Patients with mental illnesscannot sign informed consent on their own.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Interstitial lung disease and respiratory sleep apnoea
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
imaging changes and ROSE and NGS in patients | 2Day
  Relationship between imaging changes and ROSE and NGS in patients with interstitial lung disease

SECONDARY OUTCOMES:
Severity and biological examination of OSA patients | 2Day
  Classification of the severity of OSA and the relationship between positive results of biological or other tests

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China